CLINICAL TRIAL: NCT02167425
Title: Reducing Failure-to-Initiate ART Among People Who Inject Drugs: the IMAT Strategy
Brief Title: Study of Integrating Antiretroviral Therapy With Methadone Treatment for People Who Inject Drugs
Acronym: IMAT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Pangaea Global AIDS Foundation (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IMAT-01; R34DA037787 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: HIV; Opioid Dependence
Keywords: People who Inject Drugs; HIV; Methadone; Sub Saharan Africa; Tanzania; Implementation Science
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Late Post-IMAT Cohort: Enrollment into the Late Post-IMAT Cohort will occur over a 9-month period in beginning in the second year of the intervention and will be followed by a 3-month period of follow-up after the close of enrollment.
  Interventions: Other: IMAT
- Early Post-IMAT Cohort: Enrollment into the Early Post-IMAT Cohort will occur over a 9-month period immediately following the intervention and will be followed by a 3-month period of follow-up after the close of enrollment.
  Interventions: Other: IMAT
- Late Pre-IMAT Cohort: Enrollment into the Late Pre-IMAT Cohort will begin one year prior to implementation of the intervention. Enrollment will occur over a 9-month period and will be followed by a 3-month period of follow-up after the close of enrollment.
- Early Pre-IMAT Cohort: Enrollment into the Early Pre-IMAT Cohort will begin two years prior to implementation of the intervention. Enrollment will occur over a 9-month period and will be followed by a 3-month period of follow-up after the close of enrollment.

INTERVENTIONS:
Other: IMAT — The IMAT intervention will combine three main strategies: point-of-care (POC) CD4 screening, provider training and mentoring, and an alerts and reminder dashboard. The POC CD4 platform will provide real-time clinical staging, enabling providers within the methadone clinic to screen HIV-infected patients for ART eligibility. Coupled with this technology, appropriate training and mentoring will predispose providers to effectively link patients to ART and integration of an alert and reminder dashboard will reinforce behavior change and strengthen processes.
  Other Names: Integrated Methadone and Antiretroviral Therapy
  Groups: Early Post-IMAT Cohort; Late Post-IMAT Cohort

SUMMARY:
To improve ART initiation among people who inject drugs, the investigators propose to develop and pilot a multi-component Integrated Methadone and Antiretroviral Therapy strategy (IMAT) in Dar es Salaam, Tanzania. In doing so, the investigators anticipate building a functional model of methadone and ART integration that improves the effectiveness and efficiency of service delivery.

DETAILED DESCRIPTION:
The overarching goal of the proposed research is to develop and test an innovative implementation model (IMAT) for the effective integration of HIV care and treatment with methadone services in Dar es Salaam, Tanzania. The investigators will utilize the PRECEDE framework to inform the intervention to improve linkage of HIV-positive methadone patients to ART. This model suggests that strategies intended to improve health care delivery should consider a combination of three factors: 1) 'predisposing factors' - characteristics such as knowledge, attitudes, beliefs and motivation to change, 2) 'enabling factors' - characteristics that enable someone to act on their desired behavior and 3) 'reinforcing factors' - factors that encourage repetition or persistence of behavior. Therefore, our IMAT approach uses 1) targeted education and mentoring for providers that predispose them to timely ART initiation, 2) POC CD4 count platforms (PIMA, Alere) providing real-time screening and results that enable ART initiation and 3) an alerts and reminder dashboard (e.g., a summary of key indicators for improved decision making) for providers that reinforce ART initiation. Additionally, our approach will lay the foundation for developing implementation strategies for future point-of-care technologies such as viral load.

The study will combine a mixture of qualitative and quantitative methodologies to inform and evaluate the IMAT intervention.

A baseline qualitative study using in-depth interviews will be conducted among providers and methadone clients to understand predisposing, enabling and reinforcing factors related to integration of HIV care and treatment into the methadone clinic. Information gained from these qualitative assessments will inform and support the IMAT strategy. In addition, HIV-positive methadone clients will be randomly selected to complete a baseline cross-sectional survey to collect data on patient satisfaction, access to HIV care, current treatment navigation access, and HIV care literacy.

The investigators will assess the effectiveness of IMAT with a quasi-experimental pre-post cohort design and a pre-post cross-sectional survey to examine changes in patient- and provider-level outcomes after implementation of IMAT compared to before IMAT. In addition, The investigators will assess the feasibility and acceptability of the IMAT strategy using a post-implementation cross-sectional survey with a particular emphasis on satisfaction with services; a time motion study to understand the timeliness of care provision; and in-depth interviews with patients and providers to understand experiences with the IMAT strategy.

ELIGIBILITY:
Inclusion Criteria:

Methadone clients living with HIV but not linked to ART are the primary study population. Inclusion criteria for methadone initiation:

1. opioid dependence
2. positive urine screening for opiates.

   Additional inclusion criteria include:
3. age ≥ 18 years of age
4. HIV-positive. Individuals must also be willing to provide informed consent and be fluent in Kiswahili or English to participate in cross-sectional surveys and in-depth interviews

Exclusion Criteria:

We will exclude methadone clients from this study who have

1. received ART prior to methadone initiation
2. received a tuberculosis-positive diagnosis
3. women who are pregnant. The investigators have excluded clients who have received ART in the past as their inclusion would bias our study results. The investigators have also excluded patients with a tuberculosis diagnosis or women who are pregnant as they have a unique and urgent need for treatment and should be initiated onto ART regardless of their CD4 count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sites will include the methadone clinics at Muhimbili National Hospital, Mwananyamala Regional Hospital, and Temeke Regional Hospital. The study population includes methadone patients and the providers of clinical services at these facilities.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Time to CD4 Screening | Up to 36 months
  Number of days between positive HIV test and CD4 screening. Extracted from routine clinical and laboratory monitoring data.

SECONDARY OUTCOMES:
Provider Time to Ordering CD4 Screening | Up to 36 months
  Collected via routine, programmatic data
Percentage of clients that receive CD4 screening within 30 days of HIV-positive test | Up to 36 months
  Collected via routine, programmatic data
Percentage of eligible (CD4<350) clients that initiate ART within 30 days of CD4 screening | Up to 36 months
  Collected via routine, programmatic data
Percentage of clients on ART that receive at least 95% ART doses (i.e., adherence) | Up to 36 months
  Collected via routine, programmatic data
Percentage of patients receiving HIV treatment navigation counseling from provider | Three months pre-intervention and three months post-intervention
  Collected via cross-sectional surveys pre- and post-intervention.
Percentage of patients literate in CD4 screening process | Three months pre-intervention and three months post-intervention
  Collected via cross-sectional surveys pre- and post-intervention.
Percentage of patients literate in ART Initiation process | Three months pre-intervention and three months post-intervention
  Collected via cross-sectional surveys pre- and post-intervention.
Time to ART Initiation | Up to 36 months
  Number of Days between receiving a qualifying CD4 count and first dose of ART. Extracted from routine clinical and laboratory monitoring data.

OTHER OUTCOMES:
Percentage of patients satisfied with the quality of services provided | Up to three months post-intervention
Percentage of patients satisfied with confidentiality at the facility | Up to three months post-intervention
Percentage of patients satisfied with the time services are provided | Up to three months post-intervention
Percentage of patients satisfied with waiting times | Up to three months post-intervention
Average waiting time | Up to three months post-intervention
Percentage of patients satisfied with visit times | Up to three months post-intervention
Average visit time | Up to three months post-intervention
Qualitative evaluation of feasibility and acceptability of the IMAT strategy | Up to three months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Barrot H Lambdin, PhD, MPH, Principal Investigator — Pangaea Global AIDS; Jessie Mbwambo, MD, PhD, Study Director — Muhimbili University of Health and Allied Sciences